CLINICAL TRIAL: NCT05910424
Title: Characterisation of the Oral Microbiota and Oral Status of a Population of Adult Patients With Autism Spectrum Disorders: a Pilot Study
Brief Title: Oral Microbiota and Oral Status of Adult Patients With Autism Spectrum Disorders (MICAA: MICrobiota Autism Adults)
Acronym: MICAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, BERBE Ludivine, Dentist, University Hospital Assistant, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-A01024-41
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorder; Oral microbiota; Oral Health
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Pilot study concerning adults with autism spectrum disorder
Masking Description: No Treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults with Autism Spectrum Disorder (Experimental): * Adults with autism spectrum disorder
  * Aged between 18 and 60 years old
  * Dental cares and follow-up in Nancy hospital
  Interventions: Other: collection of saliva, gum fluid and/or dental plaque samples

INTERVENTIONS:
Other: collection of saliva, gum fluid and/or dental plaque samples — Non-invasive sampling of dental plaque, crevicular fluid and/or saliva, using an examination probe, paper tips and saliva swabs

SUMMARY:
The goals of this pilot study are to assess the presence of harmful germs for gums and to assess oral health in adults with autism spectrum disorder.

DETAILED DESCRIPTION:
Participants or their tutors will fulfill a form with general health information and daily habits.

Investigators will :

* collect saliva, gum fluid and/ or dental plaque to characterise germs
* assess gum health and oral hygiene
* register decays, filled and missing teeth.

ELIGIBILITY:
Inclusion Criteria:

* A person (or legal representative) who has received full information about the organisation of the research and accept to participate and the use of his or her data.
* Adult with autism spectrum disorder, men or women aged between 18 and 60.
* Member of a social security scheme or beneficiary of a medical insurance

Exclusion Criteria:

* Children under 18 with autism spectrum disorder
* Use of medication or situations that may affect the microbiota (use of antibiotics, probiotics, steroidal or non-steroidal anti-inflammatory drugs in the last 3 months, strict mouth breathing)
* Smoking
* Very lingual position of the teeth hindering clinical assessment of the periodontium
* Patients who have had periodontal treatment for less than 6 months
* Persons covered by articles L. 1121-5 to L. 1121-7 and L1122-2 of the French Public Health Code:
* Pregnant women, women in labour or breast-feeding mothers
* Persons deprived of their liberty by a judicial or administrative decision
* Persons unable to give their consent
* Person under psychiatric care by virtue of articles L. 3212-1 and L. 3213-1 of the Public Health Code
* Minor (not emancipated)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Presence of periodontopathogenic bacteria (harmful for gums) | Collection on Day 1
  Technique used = Polymerase Chain Reaction (PCR) Measure unit = Colony-Forming Unit (CFU)

SECONDARY OUTCOMES:
Assessment of the presence of parasites Entamoeba gingivalis subtype 1 (ST1) and subtype 2 (ST2) and Trichomonas tenax | Collection on Day 1
  Technique = Polymerase Chain Reaction (PCR) Unit = Colony-Forming Unit (CFU)
Assessment of the periodontal status of patients with Autism Spectrum Disorder | Day 1
  Index used = the Dutch Periodontal Index 0 = minimum value, better outcome 4 = maximum value, worse outcome
Assessment of the dental condition | Day 1
  Dental data will be collected using the Decay-Missing-Filled/Teeth (DMFT) score 0 = minimum value, best outcome 28 = maximum value, worst outcome
Assessment of oral hygiene | Day 1
  Oral hygiene will be assessed using the Silness and Löe plaque index and the lifestyle questionnaire 0 = minimum value, best outcome 3 = maximum value, worst outcome
Collection of data about lifestyle habits (oral and dental hygiene, diet, activity, etc.) and drug treatments that may influence the clinical parameters observed | Before samples collection and clinical examination
  Data collection via a form fulfilled by the participant or the patient's legal guardian

CONTACTS AND LOCATIONS:
Overall Officials: Ludivine BERBE, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU Brabois, Vandœuvre-lès-Nancy, France